CLINICAL TRIAL: NCT04309500
Title: Development of Culturally-Sensitive and Patient-Centered Feedback for Alzheimer's Dementia Risk Disclosure
Brief Title: SHARE(D) Stage II: Alzheimer's Risk Disclosure Protocol Piloting
Acronym: SHARE(D)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Annalise Rahman-Filipiak, Assistant Professor, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00178869; 1R03AG063222-01 (NIH)
Record Dates: First submitted 2020-03-10; First posted 2020-03-16 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-01

CONDITIONS: Mild Cognitive Impairment; Healthy Aging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Stage II will involve a clinical trial, with the risk disclosure feedback serving as the behavioral intervention. The study will use a single-group design with no control group. All 10 participant-co-participant dyads (5 Non-Hispanic African-American, 5 Non-Hispanic White) will receive feedback about the participant's DAT risk. Outcomes will be measured immediately following feedback and at 1- and 6-weeks following risk disclosure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Amyloid Positive (Tau Positive or Negative) Participants (Experimental): Participants who receive results of elevated amyloid (whether or not tau is also elevated), indicating the presence of Alzheimer's disease brain changes.
  Interventions: Behavioral: Personalized DAT Risk Disclosure Protocol
- Amyloid Negative (Tau Positive or Negative) Participants (Experimental): Participants who receive results of not-elevated amyloid (whether or not tau is elevated), indicating the absence of Alzheimer's disease brain changes.
  Interventions: Behavioral: Personalized DAT Risk Disclosure Protocol
- Co-Participants of Amyloid Positive (Tau Positive or Negative) Participants (Experimental): Study partners of participants who receive results of elevated amyloid (whether or not tau is also elevated), indicating the presence of Alzheimer's disease brain changes.
  Interventions: Behavioral: Personalized DAT Risk Disclosure Protocol
- Co-Participants of Amyloid Negative (Tau Positive or Negative) Participants (Experimental): Study partners of participants who receive results of not-elevated amyloid (whether or not tau is elevated), indicating the absence of Alzheimer's disease brain changes.
  Interventions: Behavioral: Personalized DAT Risk Disclosure Protocol

INTERVENTIONS:
Behavioral: Personalized DAT Risk Disclosure Protocol — Individual participants and their co-participants will receive information about the participant's DAT risk based on their clinical history, structural magnetic resonance imaging, apolipoprotein-E (APO-E) genotype, and amyloid and tau burden on positron emission tomography (PET) scanning. This session will include consent, psychoeducation, re-consent, personal risk feedback, action suggestions, participant/caregiver resources, and a written summary of results. Risk assessment and safety planning will be applied if needed.

SUMMARY:
The goal of this study is to test efficacy and safety of person-centered, culturally-informed protocols for disclosure of different combinations of Alzheimer's dementia risk factors. Building on the results from a federally-funded assessment of preferences and needs of racially diverse participants and their respective friends/family members, in regard to Dementia - Alzheimer's Type (DAT), we have produced protocols for communication of DAT risk, with attention to specific adaptations in style or content based on individual factors and preferences. These protocols allow for communication of risk based on clinical history and diagnosis, structural neuroimaging, apolipoprotein-E status, and amyloid and tau burden on positron emission tomography. In particular, protocols specify (a) effective methods of communicating risk conferred by each data source, (b) information designed for patients versus informants, (c) psychoeducation needs, and (d) resource/support needs. We will recruit a randomly-selected subset of 10 dyads (including 5 participants who are Non-Hispanic African-American, 5 participants who are Non-Hispanic White) from the Stage I sample to whom we will develop and implement personalized DAT risk disclosure protocols. We will provide preliminary information on the effectiveness of these protocols in terms of patient/co-participant comprehension and recall of feedback provided, and initial changes in mood or behavior immediately following and shortly after risk disclosure sessions.

DETAILED DESCRIPTION:
Currently, a divide exists between Dementia - Alzheimer's Type (DAT) risk information that is shared in clinical settings versus genetic and biomarker-based risk information gathered and, less frequently, disseminated in research settings. Clinical feedback continues to discuss DAT risk in terms of personal/family history, neuropsychological or neurological testing, and standard neuroimaging reports. Research advances in genotyping, quantitative neuroimaging, and amyloid and tau positron emission tomography (PET) have improved our risk prediction and disease staging; however, the literature on how to share these important findings is sparse. Effective risk disclosure protocols are fundamentally dependent on the needs of recipients. However, we do not know how patients, or those tasked with current or future caregiving, decide what sources or types of risk information they want disclosed, nor their reasons for preferring certain types of information over others. Given the differences between static (e.g., family history, genotyping) and dynamic, potentially modifiable risk factors (e.g., amyloid burden), as well as varying familiarity with research-based biomarkers, it is especially important to understand how much information patients hope to receive and what they hope to do with it. This knowledge gap is particularly pertinent in minority and low-income populations given systemic challenges and cultural beliefs that may affect their psychological, physical, and financial ability to adapt to a high risk profile. Thus, understanding risk disclosure needs and preferences is a critical step in developing culturally-informed feedback protocols.

Aim 1 (accomplished during the Stage I observational Needs Assessment - HUM00160276) was to investigate the preferences and needs of racially diverse participants, and their respective informants, in regards to receiving feedback about their risk for DAT.

Aim 2 is to develop person-centered, culturally-informed protocols for disclosure of different combinations of Alzheimer's dementia risk factors. Building on the results of Aim 1, we have produced protocols for communication of DAT risk, with attention to specific adaptations in style or content based on individual factors and preferences. In particular, protocols specify (a) effective methods of communicating risk conferred by each data source, (b) information designed for patients versus informants, (c) psychoeducation needs, and (d) resource/support needs. We will recruit a randomly-selected subset of 10 dyads (including 5 participants who are Non-Hispanic African-American, 5 participants who are Non-Hispanic White) from the Stage I sample to whom we will develop and implement personalized DAT risk disclosure protocols. We will provide preliminary information on the effectiveness of these protocols in terms of patient/co-participant comprehension and recall of feedback provided, and initial changes in mood or behavior immediately following and shortly after risk disclosure sessions.

ELIGIBILITY:
Inclusion Criteria:

* age 65+ years
* Non-Hispanic Black or Non-Hispanic White race/ethnicity
* Previously participated in Stage I (observational needs assessment)
* Have completed an initial evaluation as part of the University of Michigan Memory and Aging Project (UM-MAP), Stimulation to Improve Memory (STIM) study, or the DAPPER study within the last 12 months.
* Diagnosed with normal cognition or mild cognitive impairment (MCI; single- or -multiple domain, amnestic or non-amnestic forms)
* Able to identify a co-participant who is currently the participant's caregiver, or would serve in this role in the future if needed, and well-known to the participant (known for ≥5 years and have at least weekly phone or in-person contact)
* Able to identify a co-participant who is 18+ years old.
* Able to identify a co-participant who is cognitively healthy

Exclusion Criteria:

* Current or historical neurologic disorder (e.g., Alzheimer's dementia or other neurodegenerative dementia, Parkinson's disease, seizure disorder, tumor, multiple sclerosis)
* Current or historical significant neurologic injury (e.g., significant stroke or moderate-severe head injury, defined by loss of consciousness > 5 minutes, presence of significant post-traumatic amnesia, or the need for extended hospitalization or intervention).
* Motor symptoms indicative of a neurodegenerative etiology other than Alzheimer's disease
* Severe mental illness (i.e., bipolar disorder, thought disorder, psychosis)
* Severe substance use disorder

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annalise M Rahman-Filipiak, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Medical School, Department of Psychiatry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available to other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Amyloid Positive (Tau Positive or Negative) Participants: Participants who receive results of elevated amyloid (whether or not tau is also elevated), indicating the presence of Alzheimer's disease brain changes.
  Personalized Dementia - Alzheimer's Type (DAT) Risk Disclosure Protocol: Individual participants and their co-participants will receive information about the participant's DAT risk based on their clinical history, structural magnetic resonance imaging, apolipoprotein-E (APO-E) genotype, and amyloid and tau burden on positron emission tomography (PET) scanning. This session will include consent, psychoeducation, re-consent, personal risk feedback, action suggestions, participant/caregiver resources, and a written summary of results. Risk assessment and safety planning will be applied if needed.
- Co-Participants of Amyloid Positive (Tau Positive or Negative) Participants: Study partners of participants who receive results of elevated amyloid (whether or not tau is also elevated), indicating the presence of Alzheimer's disease brain changes.
  Personalized Dementia - Alzheimer's Type (DAT) Risk Disclosure Protocol: Individual participants and their co-participants will receive information about the participant's DAT risk based on their clinical history, structural magnetic resonance imaging, apolipoprotein-E (APO-E) genotype, and amyloid and tau burden on positron emission tomography (PET) scanning. This session will include consent, psychoeducation, re-consent, personal risk feedback, action suggestions, participant/caregiver resources, and a written summary of results. Risk assessment and safety planning will be applied if needed.
Period: Overall Study
Arm/Group | Amyloid Positive (Tau Positive or Negative) Participants | Amyloid Negative (Tau Positive or Negative) Participants | Co-Participants of Amyloid Positive (Tau Positive or Negative) Participants | Co-Participants of Amyloid Negative (Tau Positive or Negative) Participants
Started | 5 | 5 | 5 | 5
Immediate | 5 | 5 | 5 | 5
1 Week Later | 5 | 5 | 5 | 5
6 Weeks Later | 4 | 5 | 4 | 5
Completed | 4 | 5 | 5 | 5
Not Completed | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amyloid Positive (Tau Positive or Negative) Participants | Amyloid Negative (Tau Positive or Negative) Participants | Co-Participants of Amyloid Positive (Tau Positive or Negative) Participants | Co-Participants of Amyloid Negative (Tau Positive or Negative) Participants | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.00 (5.15) | 72.60 (5.41) | 69.80 (5.54) | 75.40 (10.50) | 73.20 (6.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 4 | 11
  Male | 4 | 3 | 1 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 2 | 6
  White | 4 | 3 | 4 | 3 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 5 | 5 | 20
Continuous Years of Education [Mean (Standard Deviation); unit: years] | 17.20 (3.03) | 17.80 (3.77) | 16.20 (3.03) | 17.40 (4.88) | 17.15 (3.50)
Baseline Beck Anxiety Inventory (BAI) [Mean (Standard Deviation); unit: score on a scale] — A 21-item measure of the perceived severity ('not at all' to 'severely') at which the participant is experiencing anxiety symptoms over the past week, validated for use with older adults. The range of the scores is 0-63, with higher scores meaning greater anxiety.
  score on a scale | 2.20 (2.95) | 2.00 (3.08) | 4.40 (4.56) | 2.00 (2.55) | 2.65 (3.27)
Baseline Geriatric Depression Scale (GDS) [Mean (Standard Deviation); unit: score on a scale] — A 15-item assessment of depressive symptoms that has been adapted to remove common depression symptoms often conflated with normal aging (i.e., somatic symptoms). It asks the participant to rate the presence of mood symptoms over the past two weeks. Scores on the adapted assessment range from 0-15, with higher scores indicating more depressive symptoms.
  score on a scale | 0.80 (0.84) | 1.40 (0.89) | 0.60 (1.34) | 0.40 (0.55) | 0.80 (0.95)

OUTCOME MEASURES:

1. Primary Outcome: Comprehension/Recall of Results - Personal Information Score - PARTICIPANT
Description: Participants were asked a series of multiple choice and true/false questions about their understanding or memory of the participant's current diagnosis, structural neuroimaging, APO-E genotype, and amyloid and/or tau positivity. Scores were on a range of 0 - 100 percent correct.
Time Frame: Administered immediately after risk disclosure, at 1 week, and at 6 weeks after disclosure
Population: 1 participant in the "Amyloid Positive" arm completed the immediately after disclosure and 1-week follow-up sessions but was lost to follow-up prior to the 6-week session.
Measure: Mean (Standard Deviation); unit: percentage correct
Arm/Group | Amyloid Positive (Tau Positive or Negative) Participants | Amyloid Negative (Tau Positive or Negative) Participants
Number analyzed (Participants) | 5 | 5
percentage correct
  immediately after disclosure | 82.40 (25.07) | 94.60 (5.51)
  1 week after disclosure | 69.40 (27.73) | 90.80 (5.76)
  6 weeks after disclosure: number analyzed (Participants) | 4 | 5
  6 weeks after disclosure | 70.00 (33.56) | 90.60 (5.94)

2. Primary Outcome: Comprehension/Recall of Results - Personal Information Score - CO-PARTICIPANTS
Description: Co-participants were asked a series of multiple choice and true/false questions about their understanding or memory of the participant's current diagnosis, structural neuroimaging, APO-E genotype, and amyloid and/or tau positivity. Scores were on a range of 0 - 100 percent correct.
Time Frame: Administered immediately after risk disclosure, at 1 week, and at 6 weeks after disclosure
Population: 1 study partner in the "Co-Participants of Amyloid Positive" arm did not complete the 6-week evaluation.
Measure: Mean (Standard Deviation); unit: percentage correct
Arm/Group | Co-Participants of Amyloid Positive (Tau Positive or Negative) Participants | Co-Participants of Amyloid Negative (Tau Positive or Negative) Participants
Number analyzed (Participants) | 5 | 5
percentage correct
  immediately after disclosure | 91.60 (12.26) | 96.00 (5.87)
  1 week after disclosure | 93.20 (11.69) | 92.00 (10.95)
  6 weeks after disclosure: number analyzed (Participants) | 4 | 5
  6 weeks after disclosure | 86.00 (10.23) | 85.20 (10.69)

3. Primary Outcome: Comprehension/Recall of Results - Meaning of Risk Information Score - PARTICIPANTS
Description: Participants were asked a series of multiple choice and true/false questions about their understanding or memory of the meaning of the participant's current diagnosis, structural neuroimaging, APO-E genotype, and amyloid and/or tau positivity (i.e., whether their profile on each of these indicators was related to increased, decreased, or unclear risk for DAT). Scores were on a range of 0 - 100 percent correct.
Time Frame: Administered immediately after risk disclosure, at 1 week, and at 6 weeks after disclosure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage correct
Arm/Group | Amyloid Positive (Tau Positive or Negative) Participants | Amyloid Negative (Tau Positive or Negative) Participants
Number analyzed (Participants) | 5 | 5
percentage correct
  immediately after disclosure | 80.00 (29.92) | 83.40 (15.50)
  1 week after disclosure | 68.20 (33.72) | 88.40 (16.13)
  6 weeks after disclosure: number analyzed (Participants) | 4 | 5
  6 weeks after disclosure | 81.25 (37.50) | 90.00 (22.36)

4. Primary Outcome: Comprehension/Recall of Results - Meaning of Risk Information Score - CO-PARTICIPANTS
Description: Co-participants were asked a series of multiple choice and true/false questions about their understanding or memory of the meaning of the participant's current diagnosis, structural neuroimaging, APO-E genotype, and amyloid and/or tau positivity (i.e., whether their profile on each of these indicators was related to increased, decreased, or unclear risk for DAT). Scores were on a range of 0 - 100 percent correct.
Time Frame: Administered immediately after risk disclosure, at 1 week, and at 6 weeks after disclosure
Population: 1 study partner in the "Co-Participants of Amyloid Positive" arm did not complete the 6-week evaluation.
Measure: Mean (Standard Deviation); unit: percentage correct
Arm/Group | Co-Participants of Amyloid Positive (Tau Positive or Negative) Participants | Co-Participants of Amyloid Negative (Tau Positive or Negative) Participants
Number analyzed (Participants) | 5 | 5
percentage correct
  immediately after disclosure | 95.00 (11.18) | 68.40 (20.74)
  1 week after disclosure | 93.40 (14.76) | 68.40 (20.74)
  6 weeks after disclosure: number analyzed (Participants) | 4 | 5
  6 weeks after disclosure | 100.00 (0.00) | 63.40 (28.02)

5. Primary Outcome: Geriatric Depression Scale - Short Form (GDS-15) - PARTICIPANTS
Description: A 15-item assessment of depressive symptoms that was adapted to remove common depression symptoms often conflated with normal aging (i.e., somatic symptoms).Participant were asked to rate the presence of mood symptoms over the past two weeks. Scores for the assessment ranged from 0-15, with higher scores indicating more depressive symptoms
Time Frame: Administered immediately after risk disclosure, at 1 week, and at 6 weeks after disclosure
Population: GDS was erroneously not collected for 1 participant in each arm at the immediate and 1-week time point. 1 participant in the "Amyloid Positive" arm completed the immediately after disclosure and 1-week follow-up sessions but was lost to follow-up prior to the 6-week session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Amyloid Positive (Tau Positive or Negative) Participants | Amyloid Negative (Tau Positive or Negative) Participants
Number analyzed (Participants) | 5 | 5
score on a scale
  immediately after disclosure: number analyzed (Participants) | 4 | 4
  immediately after disclosure | 2.50 (0.58) | 1.75 (0.96)
  1 week after disclosure: number analyzed (Participants) | 4 | 4
  1 week after disclosure | 1.50 (0.58) | 2.25 (1.50)
  6 weeks after disclosure: number analyzed (Participants) | 4 | 5
  6 weeks after disclosure | 2.25 (2.06) | 1.60 (1.82)

6. Primary Outcome: Geriatric Depression Scale - Short Form (GDS-15) - CO-PARTICIPANTS
Description: A 15-item assessment of depressive symptoms that was adapted to remove common depression symptoms often conflated with normal aging (i.e., somatic symptoms). Co-participant were asked to rate the presence of mood symptoms over the past two weeks. Scores for the assessment ranged from 0-15, with higher scores indicating more depressive symptoms
Time Frame: Administered immediately after risk disclosure, at 1 week, and at 6 weeks after disclosure
Population: GDS was erroneously not collected for 1 study partner in each arm at the immediate and 1-week time point. 1 study partner in the "Co-Participants of Amyloid Positive" arm did not complete the 6-week follow-up, as it fell outside of the study funding period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Co-Participants of Amyloid Positive (Tau Positive or Negative) Participants | Co-Participants of Amyloid Negative (Tau Positive or Negative) Participants
Number analyzed (Participants) | 5 | 5
score on a scale
  immediately after disclosure: number analyzed (Participants) | 4 | 4
  immediately after disclosure | 0.25 (0.50) | 0.00 (0.00)
  1 week after disclosure: number analyzed (Participants) | 4 | 4
  1 week after disclosure | 0.75 (1.50) | 0.25 (0.50)
  6 weeks after disclosure: number analyzed (Participants) | 4 | 5
  6 weeks after disclosure | 0.75 (0.96) | 0.40 (0.89)

7. Primary Outcome: Beck Anxiety Inventory (BAI) - PARTICIPANTS
Description: A 21-item measure of the perceived severity ('not at all' to 'severely') at which the participant was experiencing anxiety symptoms over the past week, validated for use with older adults. Scores ranged from 0-63, with higher scores indicating greater anxiety.
Time Frame: Administered immediately after risk disclosure, at 1 week, and at 6 weeks after disclosure
Population: BAI was erroneously not collected for 1 participant in each arm at the immediate and 1-week time point. 1 participant in the "Amyloid Positive" arm completed the immediately after disclosure and 1-week follow-up sessions but was lost to follow-up prior to the 6-week session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Amyloid Positive (Tau Positive or Negative) Participants | Amyloid Negative (Tau Positive or Negative) Participants
Number analyzed (Participants) | 5 | 5
score on a scale
  immediately after disclosure: number analyzed (Participants) | 4 | 4
  immediately after disclosure | 6.75 (8.06) | 2.25 (4.50)
  1 week after disclosure: number analyzed (Participants) | 4 | 4
  1 week after disclosure | 0.75 (0.96) | 1.25 (1.89)
  6 weeks after disclosure: number analyzed (Participants) | 4 | 5
  6 weeks after disclosure | 0.00 (0.00) | 4.00 (5.15)

8. Primary Outcome: Beck Anxiety Inventory (BAI) - CO-PARTICIPANTS
Description: A 21-item measure of the perceived severity ('not at all' to 'severely') at which the co-participant was experiencing anxiety symptoms over the past week, validated for use with older adults. Scores ranged from 0-63, with higher scores indicating greater anxiety.
Time Frame: Administered immediately after risk disclosure, at 1 week, and at 6 weeks after disclosure
Population: BAI was erroneously not collected for 1 study partner in each arm at the immediate and 1-week time point. 1 study partner in the "Co-Participants of Amyloid Positive" arm did not complete the 6-week follow-up, as it fell outside of the study funding period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Co-Participants of Amyloid Positive (Tau Positive or Negative) Participants | Co-Participants of Amyloid Negative (Tau Positive or Negative) Participants
Number analyzed (Participants) | 5 | 5
score on a scale
  immediately after disclosure: number analyzed (Participants) | 4 | 4
  immediately after disclosure | 1.75 (2.22) | 1.00 (0.82)
  1 week after disclosure: number analyzed (Participants) | 4 | 4
  1 week after disclosure | 3.50 (6.35) | 0.00 (0.00)
  6 weeks after disclosure: number analyzed (Participants) | 4 | 5
  6 weeks after disclosure | 5.25 (6.08) | 1.20 (1.64)

9. Primary Outcome: The Impact of Genetic Testing for AD (IGT-AD; Positive Subscale) - PARTICIPANTS
Description: The Impact of Genetic Testing for AD (IGT-AD) (positive subscale) was a 4-item self-report measure that assessed two positive and negative emotional responses to genetic AD risk disclosure. This scale was adapted to more broadly assess the 'life event' of receiving DAT risk disclosure based on multiple indicators. Participants completed this to assess their reactions to the participant receiving risk feedback. Possible scores ranged from 0 - 60, where 0 meant fewest positive reactions and 20 was most (strongest) positive reactions.
Time Frame: Administered immediately after risk disclosure, at 1 week, and at 6 weeks after disclosure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Amyloid Positive (Tau Positive or Negative) Participants | Amyloid Negative (Tau Positive or Negative) Participants
Number analyzed (Participants) | 5 | 5
score on a scale
  immediately after disclosure | 14.20 (5.59) | 16.80 (4.15)
  1 week after disclosure | 14.50 (5.97) | 18.40 (2.61)
  6 weeks after disclosure: number analyzed (Participants) | 4 | 5
  6 weeks after disclosure | 9.75 (5.19) | 18.40 (2.19)

10. Primary Outcome: The Impact of Genetic Testing for AD (IGT-AD; Positive Subscale) - CO-PARTICIPANTS
Description: The Impact of Genetic Testing for AD (IGT-AD) (positive subscale) was a 4-item self-report measure that assessed two positive and negative emotional responses to genetic AD risk disclosure. This scale was adapted to more broadly assess the 'life event' of receiving DAT risk disclosure based on multiple indicators. Co-participants completed this to assess their reactions to the participant receiving risk feedback. Scores ranged from 0 - 60, where 0 meant fewest positive reactions and 20 was most (strongest) positive reactions.
Time Frame: Administered immediately after risk disclosure, at 1 week, and at 6 weeks after disclosure
Population: One study partner in the "Co-Participants of Amyloid Positive" arm did not complete the 6-week follow-up as it fell outside of the study funding period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Co-Participants of Amyloid Positive (Tau Positive or Negative) Participants | Co-Participants of Amyloid Negative (Tau Positive or Negative) Participants
Number analyzed (Participants) | 5 | 5
score on a scale
  Immediately after disclosure | 17.20 (3.03) | 17.80 (3.90)
  1 week after disclosure | 10.80 (4.76) | 19.60 (0.89)
  6 weeks after disclosure: number analyzed (Participants) | 4 | 5
  6 weeks after disclosure | 10.50 (1.00) | 19.20 (1.10)

11. Primary Outcome: The Impact of Genetic Testing for AD (IGT-AD; Distress Subscale) - PARTICIPANTS
Description: The Impact of Genetic Testing for AD (IGT-AD) was a 16-item self-report measure that assessed two positive and negative emotional responses to genetic AD risk disclosure. This scale was adapted to more broadly assess the 'life event' of receiving DAT risk disclosure based on multiple indicators. Participants completed this to assess their reactions to the participant receiving risk feedback.
  The Distress subscale scores ranged from 0-60, with higher scores indicating greater distress about test results.
Time Frame: Administered immediately after risk disclosure, at 1 week, and at 6 weeks after disclosure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Amyloid Positive (Tau Positive or Negative) Participants | Amyloid Negative (Tau Positive or Negative) Participants
Number analyzed (Participants) | 5 | 5
score on a scale
  Immediately after disclosure | 13.60 (9.66) | 3.40 (3.58)
  1 week after disclosure | 5.60 (7.83) | 4.20 (2.78)
  6 weeks after disclosure: number analyzed (Participants) | 4 | 5
  6 weeks after disclosure | 5.25 (6.40) | 4.00 (5.15)

12. Primary Outcome: The Impact of Genetic Testing for AD (IGT-AD; Distress Subscale) - CO-PARTICIPANTS
Description: as for outcome 11
Time Frame: Administered immediately after risk disclosure, at 1 week, and at 6 weeks after disclosure
Population: One participant in the "Co-Participant of Amyloid Positive" arm did not complete the 6-week follow-up as it fell outside of the study funding period.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Co-Participants f Amyloid Positive (Tau Positive or Negative) Participants: Study partners of participants who receive results of elevated amyloid (whether or not tau is also elevated), indicating the presence of Alzheimer's disease brain changes.
  Personalized Dementia - Alzheimer's Type (DAT) Risk Disclosure Protocol: Individual participants and their co-participants will receive information about the participant's DAT risk based on their clinical history, structural magnetic resonance imaging, apolipoprotein-E (APO-E) genotype, and amyloid and tau burden on positron emission tomography (PET) scanning. This session will include consent, psychoeducation, re-consent, personal risk feedback, action suggestions, participant/caregiver resources, and a written summary of results. Risk assessment and safety planning will be applied if needed.
Arm/Group | Co-Participants f Amyloid Positive (Tau Positive or Negative) Participants | Co-Participants of Amyloid Negative (Tau Positive or Negative) Participants
Number analyzed (Participants) | 5 | 5
score on a scale
  Immediately after disclosure | 10.60 (11.19) | 5.40 (4.93)
  1 week after disclosure | 18.80 (14.06) | 2.60 (2.97)
  6 weeks after disclosure: number analyzed (Participants) | 4 | 5
  6 weeks after disclosure | 9.00 (9.49) | 3.00 (3.46)

13. Other Pre Specified Outcome: Comprehension of Results - Qualitative Impressions
Description: Participants and co-participants were asked to explain, in their own words and without cuing, their impressions of the messages they received about the participant's clinical history, structural neuroimaging, genetic profile, and amyloid and tau biomarkers, as well as the risk for DAT conferred by those markers. Responses were transcribed and coded to determine core themes and understanding of risk messages.
Time Frame: Administered immediately after risk disclosure; 1 week later, and 6 weeks later
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: six weeks
Arm/Group | Amyloid Positive (Tau Positive or Negative) Participants | Amyloid Negative (Tau Positive or Negative) Participants | Co-Participants of Amyloid Positive (Tau Positive or Negative) Participants | Co-Participants of Amyloid Negative (Tau Positive or Negative) Participants
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT04309500/Prot_SAP_000.pdf
  • Informed Consent Form: Consent Form - Co-Participants (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT04309500/ICF_002.pdf
  • Informed Consent Form: Consent Form - Participants (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT04309500/ICF_003.pdf